CLINICAL TRIAL: NCT01160744
Title: An Open-label, Multicenter, Randomized, Phase 2 Study of a Recombinant Human Anti-VEGFR-2 Monoclonal Antibody, IMC-1121B in Combination With Platinum-based Chemotherapy Versus Platinum-based Chemotherapy Alone as First-line Treatment of Patients With Recurrent or Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Pemetrexed and Carboplatin/Cisplatin or Gemcitabine and Carboplatin/Cisplatin With or Without IMC-1121B in Participants Previously Untreated With Recurrent or Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13916; I4T-IE-JVBL (Other: Eli Lilly and Company); CP12-0917 (Other: ImClone Systems); 2009-016784-11 (EudraCT Number)
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Results first posted 2014-12-29 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung neoplasms; Lung cancer; Non-small Cell Lung Cancer; pemetrexed; squamous; nonsquamous
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Ramucirumab; Pemetrexed; Carboplatin; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IMC-1121B + Pemetrexed + Carboplatin (AUC 6) or Cisplatin (Experimental): IMC-1121B + Pemetrexed + Carboplatin [Area Under the Concentration Time Curve 6 (AUC 6)] or Cisplatin
  Interventions: Biological: IMC-1121B (ramucirumab); Drug: Pemetrexed; Drug: Carboplatin (AUC 6); Drug: Cisplatin
- Pemetrexed + Carboplatin (AUC 6) or Cisplatin (Active Comparator): Pemetrexed + Carboplatin (AUC 6) or Cisplatin
  Interventions: Drug: Pemetrexed; Drug: Carboplatin (AUC 6); Drug: Cisplatin
- IMC-1121B + Gemcitabine + Carboplatin (AUC 5) or Cisplatin (Experimental): IMC-1121B + Gemcitabine + Carboplatin [Area Under the Concentration Time Curve 5 (AUC 5)] or Cisplatin
  Interventions: Biological: IMC-1121B (ramucirumab); Drug: Cisplatin; Drug: Gemcitabine; Drug: Carboplatin (AUC 5)
- Gemcitabine + Carboplatin (AUC 5) or Cisplatin (Active Comparator): Gemcitabine + Carboplatin (AUC 5) or Cisplatin
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Carboplatin (AUC 5)

INTERVENTIONS:
Biological: IMC-1121B (ramucirumab) — 10 milligrams/kilogram (mg/kg) once every 3 weeks beginning Day 1, Cycle 1
  Other Names: ramucirumab; IMC-1121B; LY3009806
  Arms: IMC-1121B + Gemcitabine + Carboplatin (AUC 5) or Cisplatin; IMC-1121B + Pemetrexed + Carboplatin (AUC 6) or Cisplatin
Drug: Pemetrexed — 500 milligrams/square meter (mg/m²) on Day 1 of every 21-day cycle
  Arms: IMC-1121B + Pemetrexed + Carboplatin (AUC 6) or Cisplatin; Pemetrexed + Carboplatin (AUC 6) or Cisplatin
Drug: Carboplatin (AUC 6) — Day 1 of every 21-day cycle
  Arms: IMC-1121B + Pemetrexed + Carboplatin (AUC 6) or Cisplatin; Pemetrexed + Carboplatin (AUC 6) or Cisplatin
Drug: Cisplatin — 75 mg/m² intravenous (IV) on Day 1 of each 21-day cycle
Drug: Gemcitabine — 1000 mg/m² on Days 1 and 8 of every 21-day cycle
  Arms: Gemcitabine + Carboplatin (AUC 5) or Cisplatin; IMC-1121B + Gemcitabine + Carboplatin (AUC 5) or Cisplatin
Drug: Carboplatin (AUC 5) — Day 1 of every 21-day cycle
  Arms: Gemcitabine + Carboplatin (AUC 5) or Cisplatin; IMC-1121B + Gemcitabine + Carboplatin (AUC 5) or Cisplatin

SUMMARY:
The purpose of this study is to determine if participants with Stage IV NSCLC have a better outcome when treated with IMC-1121B in combination with pemetrexed + carboplatin/cisplatin or gemcitabine + carboplatin/cisplatin than when treated with pemetrexed + carboplatin/cisplatin or gemcitabine + carboplatin/cisplatin alone.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed NSCLC
* Stage IV disease at the time of study entry
* Measurable disease at the time of study entry
* Resolution to Grade ≤ 1 Adverse Events, of all clinically significant toxic effects of prior chemotherapy, surgery, radiotherapy, or hormonal therapy (except alopecia)
* Adequate hematologic function, hepatic function, renal function and coagulation function
* If sexually active, must be post-menopausal, surgically sterile, or using effective contraception; and agrees to use adequate contraception during the study period and for up to 6 months after the last dose of study medication
* Female participants of childbearing potential must have a negative serum pregnancy test

Exclusion Criteria:

* Has cirrhosis at a level of Child-Pugh B (or worse), or cirrhosis and a history of hepatic encephalopathy, or ascites resulting from cirrhosis and requiring ongoing treatment with diuretics and/or paracentesis
* Tumor wholly or partially contains small cell lung cancer
* Untreated central nervous system (CNS) metastases, eligible if they are clinically stable with regard to neurologic function, off all steroids after cranial irradiation at least 2 weeks prior or after surgical resection performed at least 4 weeks prior to randomization
* Concurrent active malignancy other than adequately treated basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix. A participant with previous history of malignancy other than NSCLC is eligible, provided that he/she has been free of disease for ≥ 3 years
* Received prior therapy with monoclonal antibodies, signal transduction inhibitors, or any therapies targeting the vascular endothelial growth factor (VEGF) or vascular endothelial growth factor receptor (VEGFR)
* Receiving concurrent treatment with other anticancer therapy
* Has received previous chemotherapy for Stage IV NSCLC (participants who have received adjuvant chemotherapy are eligible if the last administration of the prior adjuvant regimen occurred at least 6 months prior to randomization)
* Has radiologically documented evidence of major blood vessel invasion or encasement by cancer
* Has undergone chest irradiation within 12 weeks prior to randomization (except palliative irradiation of bone lesions)
* Ongoing or active infection
* History of significant neurological or psychiatric disorders
* Experienced clinically relevant coronary artery disease, myocardial infarction within 6 months prior to randomization, uncontrolled congestive heart failure, or symptomatic poorly controlled arrhythmia
* Poorly-controlled hypertension
* Experienced any serious Grade 3-4 gastrointestinal bleeding within 3 months prior to study entry
* Receiving chronic daily treatment with aspirin (> 325 mg/day) or other known inhibitors of platelet function
* Serious nonhealing wound, ulcer, or bone fracture within 28 days prior to randomization
* Major surgery within 28 days prior the first dose of study medication, or subcutaneous venous access device placement within 7 days prior to randomization
* Elective or a planned major surgery
* Pregnant or lactating
* Any other serious uncontrolled medical disorders or psychological conditions
* Allergy / history of hypersensitivity reaction to any of the treatment components
* History of drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2010-09; Primary Completion 2014-01 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (53):
- United States (38):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corona, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fountain Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riverside, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alexandria, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lincoln, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neptune City, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Latham, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Bronx, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Langhorne, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hilton Head Island, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bedford, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., El Paso, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Worth, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kerrville, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Longview, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., McAllen, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Midland, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Woodlands, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tyler, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waco, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Christiansburg, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fairfax, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane Valley, Washington
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent, Belgium
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erlangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Großhansdorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hemer
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Karlsruhe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Regensburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
- Poland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olsztyn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- United Kingdom (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangor, Gwynedo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Doebele RC, Spigel D, Tehfe M, Thomas S, Reck M, Verma S, Eakle J, Bustin F, Goldschmidt J Jr, Cao D, Alexandris E, Yurasov S, Camidge DR, Bonomi P. Phase 2, randomized, open-label study of ramucirumab in combination with first-line pemetrexed and platinum chemotherapy in patients with nonsquamous, advanced/metastatic non-small cell lung cancer. Cancer. 2015 Mar 15;121(6):883-92. doi: 10.1002/cncr.29132. Epub 2014 Nov 6. PMID 25377507

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who died (any cause) or had disease progression were considered to be study completers.
Groups:
- Pem + Carb or Cis (Non-Squamous): Pemetrexed (Pem): 500 milligrams/square meter (mg/m²) on Day 1 of every 21-day cycle.
  Carboplatin (Carb) [Area Under the Concentration Time Curve 6 (AUC 6)] : Day 1 of every 21-day cycle.
  Cisplatin (Cis): 75 mg/m² intravenous (IV) on Day 1 of every 21-day cycle. Participants were treated for up to 89 weeks.
- Ram + Pem + Carb or Cis (Non-Squamous): Ramucirumab (Ram): 10 milligrams/kilogram (mg/kg) Day 1 of every 21-day cycle. Pem: 500 mg/m² on Day 1 of every 21-day cycle. Carb (AUC 6): Day 1 of every 21-day cycle. Cis: 75 mg/m² IV on Day 1 of every 21-day cycle. Participants were treated for up to 89 weeks.
- Gem + Carb or Cis (Squamous): Gemcitabine (Gem): 1000 mg/m² on Days 1 and 8 of every 21-day cycle. Carb [Area Under the Concentration Time Curve 5 (AUC 5)]: Day 1 of every 21-day cycle.
  Cis: 75 mg/m² IV on Day 1 of every 21-day cycle. Participants were treated for up to 89 weeks.
- Ram + Gem + Carb or Cis (Squamous): Ram: 10 mg/kg on Day 1 of each every 21-day cycle. Gem: 1000 mg/m² on Days 1 and 8 of every 21-day cycle. Carb (AUC 5): Day 1 of every 21-day cycle. Cis: 75 mg/m² IV on Day 1 of each every 21-day cycle. Participants were treated for up to 89 weeks.
Period: Overall Study
Arm/Group | Pem + Carb or Cis (Non-Squamous) | Ram + Pem + Carb or Cis (Non-Squamous) | Gem + Carb or Cis (Squamous) | Ram + Gem + Carb or Cis (Squamous)
Started | 71 | 69 | 69 | 71
Received Study Drug | 69 | 67 | 63 | 71
Completed | 60 | 64 | 62 | 67
Not Completed | 11 | 5 | 7 | 4
Not completed — Withdrawal by Subject | 11 | 5 | 6 | 4
Not completed — Not meet inclusion/exclusion criteria | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Pem + Carb or Cis (Non-Squamous): Pem: 500 mg/m² on Day 1 of every 21-day cycle. Carb (AUC 6): Day 1 of every 21-day cycle. Cis: 75 mg/m² IV on Day 1 of every 21-day cycle. Participants were treated for up to 89 weeks.
- Ram + Pem + Carb or Cis (Non-Squamous): Ram: 10 mg/kg Day 1 of every 21-day cycle. Pem: 500 mg/m² on Day 1 of every 21-day cycle. Carb (AUC 6): Day 1 of every 21-day cycle. Cis: 75 mg/m² IV on Day 1 of every 21-day cycle. Participants were treated for up to 89 weeks.
- Gem + Carb or Cis (Squamous): Gem: 1000 mg/m² on Days 1 and 8 of every 21-day cycle. Carb (AUC 5): Day 1 of every 21-day cycle. Cis: 75 mg/m² IV on Day 1 of every 21-day cycle. Participants were treated for up to 89 weeks.
- Ram + Gem + Carb or Cis (Squamous): Ram: 10 mg/kg on Day 1 of each every 21-day cycle. Gem: 1000 mg/m² on Days 1 and 8 of every 21-day cycle. Carb (AUC 5): Day 1 of every 21-day cycle. Cis: 75 mg/m² IV on Day 1 of every 21-day cycle. Participants were treated for up to 89 weeks.
- Total: Total of all reporting groups
Arm/Group | Pem + Carb or Cis (Non-Squamous) | Ram + Pem + Carb or Cis (Non-Squamous) | Gem + Carb or Cis (Squamous) | Ram + Gem + Carb or Cis (Squamous) | Total
Number analyzed (Participants) | 71 | 69 | 69 | 71 | 280
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 37 | 27 | 34 | 135
  >=65 years | 34 | 32 | 40 | 37 | 143
  Missing Data | 0 | 0 | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 33 | 26 | 16 | 101
  Male | 45 | 36 | 43 | 55 | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 1 | 0 | 6
  Not Hispanic or Latino | 70 | 65 | 68 | 71 | 274
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 65 | 60 | 65 | 67 | 257
  Black | 2 | 8 | 1 | 4 | 15
  Asian | 4 | 1 | 1 | 0 | 6
  Other | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 71 | 69 | 42 | 41 | 223
  Canada | 0 | 0 | 4 | 1 | 5
  Belgium | 0 | 0 | 5 | 4 | 9
  Poland | 0 | 0 | 4 | 12 | 16
  Germany | 0 | 0 | 14 | 8 | 22
  United Kingdom | 0 | 0 | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was the time from randomization to the first objective progression as defined by Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v 1.1) or death from any cause, whichever occurred first. Progressive disease (PD) was defined as ≥20% increase in sum of diameter (SOD) of target lesions and short axes of target lymph nodes, taking as reference the smallest sum of the longest diameters recorded since treatment started and an absolute increase in sum diameter of ≥5 millimeters (mm); appearance of ≥1 new lesions and/or unequivocal progression of existing non-target lesions. Participants alive and without disease progression were censored at the time of the last objective tumor assessment. Participants who did not progress and were lost to follow-up were censored at their last radiographic assessment. If no baseline or post baseline radiologic assessments were available, participants were censored at date of randomization.
Time Frame: Randomization to PD or death (up to 24 months)
Population: Intent-to-Treat (ITT) Population: All randomized participants. Participants censored: Pem+Carb/Cis=14, Ram+Pem+Carb/Cis=13, Gem+Carb/Cis=14, Ram+Gem+Carb/Cis=18.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Pem + Carb or Cis (Non-Squamous) | Ram + Pem + Carb or Cis (Non-Squamous) | Gem + Carb or Cis (Squamous) | Ram + Gem + Carb or Cis (Squamous)
Number analyzed (Participants) | 71 | 69 | 69 | 71
months | 5.6 [4.0 to 5.7] | 7.2 [5.8 to 8.4] | 5.4 [4.7 to 5.7] | 5.6 [4.4 to 6.0]
Statistical Analysis 1: Comparison: Pem + Carb or Cis (Non-Squamous) vs Ram + Pem + Carb or Cis (Non-Squamous); Test type: Superiority or Other; p = 0.1318, Log Rank; Hazard Ratio (HR) = 0.75, 90% CI 2-sided [0.55 to 1.03]
Statistical Analysis 2: Comparison: Gem + Carb or Cis (Squamous) vs Ram + Gem + Carb or Cis (Squamous); Test type: Superiority or Other; p = 0.5215, Log Rank; Hazard Ratio (HR) = 0.88, 90% CI 2-sided [0.64 to 1.22]

2. Secondary Outcome: Percentage of Participants With Best Overall Response of Complete Response (CR) or Partial Response (PR) [Objective Response Rate (ORR)]
Description: Best overall response of CR or PR was defined using RECIST v 1.1 criteria. CR was defined as the disappearance of all lesions, pathological lymph node reduction in short axis to <10 mm, and normalization of tumor marker levels of non-target lesions. PR was defined as ≥30% decrease in SOD of target lesions taking as reference the baseline sum diameter. PD was defined as ≥20% increase in SOD of target lesions and short axes of target lymph nodes, taking as reference the smallest sum of the longest diameters recorded since treatment started and an absolute increase in sum diameter of ≥5 mm; appearance of ≥1 new lesions and/or unequivocal progression of existing non-target lesions. Participants who had no post baseline tumor assessments were considered non-responders and included in the denominator when calculating response rate. Percentage of participants=(number of participants with CR+PR/total number of participants)*100.
Time Frame: Day 1, Cycle 1 (3-week cycles) and every 6 weeks thereafter to PD (up to 24 months)
Population: ITT Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Pem + Carb or Cis (Non-Squamous) | Ram + Pem + Carb or Cis (Non-Squamous) | Gem + Carb or Cis (Squamous) | Ram + Gem + Carb or Cis (Squamous)
Number analyzed (Participants) | 71 | 69 | 69 | 71
percentage of participants | 38.0 | 49.3 | 24.6 | 46.5
Statistical Analysis 1: Comparison: Pem + Carb or Cis (Non-Squamous) vs Ram + Pem + Carb or Cis (Non-Squamous); Test type: Superiority or Other; p = 0.1797, Chi-squared; Odds Ratio (OR) = 1.58, 90% CI 2-sided [0.90 to 2.78]
Statistical Analysis 2: Comparison: Gem + Carb or Cis (Squamous) vs Ram + Gem + Carb or Cis (Squamous); Test type: Superiority or Other; p = 0.0070, Chi-squared; Odds Ratio (OR) = 2.66, 90% CI 2-sided [1.45 to 4.86]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. If the participant was alive at the end of the follow-up period or was lost to follow-up, OS was censored on the last date the participant was known to be alive.
Time Frame: Randomization to the date of death from any cause (up to 31.3 months)
Population: ITT Population: All randomized participants. Participants censored: Pem+Carb/Cis=22, Ram+Pem+Carb/Cis=16, Gem+Carb/Cis=32, Ram+Gem+Carb/Cis=32. Censored participants were included in the analysis.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Pem + Carb or Cis (Non-Squamous) | Ram + Pem + Carb or Cis (Non-Squamous) | Gem + Carb or Cis (Squamous) | Ram + Gem + Carb or Cis (Squamous)
Number analyzed (Participants) | 71 | 69 | 69 | 71
months | 10.4 [8.2 to 15.9] | 13.9 [10.0 to 17.8] | 11.3 [9.7 to 13.3] | 10.4 [7.8 to 14.8]
Statistical Analysis 1: Comparison: Pem + Carb or Cis (Non-Squamous) vs Ram + Pem + Carb or Cis (Non-Squamous); Test type: Superiority or Other; p = 0.8916, Log Rank; Hazard Ratio (HR) = 1.03, 90% CI 2-sided [0.74 to 1.42]
Statistical Analysis 2: Comparison: Gem + Carb or Cis (Squamous) vs Ram + Gem + Carb or Cis (Squamous); Test type: Superiority or Other; p = 0.6847, Log Rank; Hazard Ratio (HR) = 0.93, 90% CI 2-sided [0.68 to 1.27]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was measured from the time criteria were met for the first objectively recorded CR or PR until the first date criteria for PD were met or death. Response was defined using RECIST v 1.1 criteria. CR was defined as the disappearance of all lesions, pathological lymph node reduction in short axis to <10 mm, and normalization of tumor marker level of non-target lesions. PR was defined as ≥30% decrease SOD of target lesions taking as reference the baseline sum diameter. PD was defined as ≥20% increase in SOD of target lesions and short axes of target lymph nodes, taking as reference the smallest sum of the longest diameters recorded since treatment started and an absolute increase in sum diameter of ≥5 mm; appearance of ≥1 new lesions and/or unequivocal progression of existing non-target lesions. Participants who did not relapse were censored at the day of their last objective tumor assessment.
Time Frame: Time of first response (CR or PR) until PD or death (up to 24 months)
Population: All randomized participants with a best overall response of CR or PR. Participants censored: Pem+Carb/Cis=44, Ram+Pem+Carb/Cis=35, Gem+Carb/Cis=50, Ram+Gem+Carb/Cis=37.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Pem + Carb or Cis (Non-Squamous) | Ram + Pem + Carb or Cis (Non-Squamous) | Gem + Carb or Cis (Squamous) | Ram + Gem + Carb or Cis (Squamous)
Number analyzed (Participants) | 27 | 34 | 17 | 33
months | 4.5 [3.1 to 5.7] | 5.5 [4.4 to 5.8] | 4.3 [4.2 to 5.5] | 4.3 [3.3 to 5.6]

5. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) and Who Died
Description: Data presented are the number of participants with at least 1 treatment-emergent adverse event (TEAE) and treatment-emergent serious adverse event (SAE), as well as, the number of participants who died during the study. TEAEs were defined as serious and other non-serious AEs that occurred or worsened after study treatment (regardless of causality). A summary of SAEs and other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Day 1, Cycle 1 (3-week cycles) Up to 3 Years
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pem + Carb or Cis (Non-Squamous) | Ram + Pem + Carb or Cis (Non-Squamous) | Gem + Carb or Cis (Squamous) | Ram + Gem + Carb or Cis (Squamous)
Number analyzed (Participants) | 69 | 67 | 63 | 71
Participants
  Treatment-Emergent SAE | 38 | 44 | 29 | 39
  Treatment-Emergent Adverse Event | 68 | 67 | 63 | 71
  Deaths | 51 | 55 | 55 | 56

6. Other Pre Specified Outcome: Percentage of Participants With CR, PR, or Stable Disease (SD) [Disease Control Rate (DCR)]
Description: DCR: percentage of participants with CR, PR, or SD using RECIST v 1.1 criteria. CR: disappearance of all lesions, pathological lymph node reduction in short axis to <10 mm, and normalization of tumor marker levels of non-target lesions. PR: ≥30% decrease in SOD of target lesions taking as reference baseline sum diameter. PD: ≥20% increase in SOD of target lesions and short axes of target lymph nodes, taking as reference smallest sum of longest diameters recorded since treatment started and an absolute increase in sum diameter ≥5 mm; appearance of ≥1 new lesions and/or unequivocal progression of existing non-target lesions. SD: neither sufficient shrinkage to qualify for PR nor increase to qualify for PD. Participants who had no post baseline tumor assessments were considered non-responders and included in the denominator when calculating response rate. Percentage of participants=(number of participants with CR+PR+SD/total number of participants)*100.
Time Frame: Day 1, Cycle 1 (3-week cycles) and every 6 weeks thereafter to PD (up to 24 months)
Population: ITT Population: All randomized participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Ram + Pem + Carb or Cis (Non-Squamous): Ram: 10 mg/kg Day 1 of every 21-day cycle. Pem: 500 mg/m² on Day 1 of every 21-day cycle. Carb (AUC 6): Day 1 of every 21-day cycle. Cisplatin: 75 mg/m² IV on Day 1 of each 21-day cycle. Participants were treated for up to 89 weeks.
- Ram + Gem + Carb or Cis (Squamous): Ram: 10 mg/kg Day 1 of every 21-day cycle. Gem: 1000 mg/m² on Days 1 and 8 of every 21-day cycle. Carb (AUC 5): Day 1 of every 21-day cycle. Cis: 75 mg/m² IV on Day 1 of every 21-day cycle. Participants were treated for up to 89 weeks.
Arm/Group | Pem + Carb or Cis (Non-Squamous) | Ram + Pem + Carb or Cis (Non-Squamous) | Gem + Carb or Cis (Squamous) | Ram + Gem + Carb or Cis (Squamous)
Number analyzed (Participants) | 71 | 69 | 69 | 71
percentage of participants | 70.4 [61.5 to 79.3] | 85.5 [78.5 to 92.5] | 66.7 [57.3 to 76.0] | 73.2 [64.6 to 81.9]
Statistical Analysis 1: Comparison: Pem + Carb or Cis (Non-Squamous) vs Ram + Pem + Carb or Cis (Non-Squamous); Test type: Superiority or Other; p = 0.0316, Chi-squared; Odds Ratio (OR) = 2.48, 90% CI 2-sided [1.22 to 5.02]
Statistical Analysis 2: Comparison: Gem + Carb or Cis (Squamous) vs Ram + Gem + Carb or Cis (Squamous); Test type: Superiority or Other; p = 0.3962, Chi-squared; Odds Ratio (OR) = 1.37, 90% CI 2-sided [0.74 to 2.52]

7. Other Pre Specified Outcome: Change in Tumor Size (CTS)
Description: CTS was defined as the log ratio of tumor size at 6 weeks to tumor size at baseline. CTS at 6 weeks=Log (Sum of Target Lesion Measurements at 6 Weeks)-Log (Sum of Target Lesion Measurements at Baseline).
Time Frame: Baseline, 6 weeks
Population: All randomized participants with results at baseline and 6 weeks.
Measure: Mean (Standard Deviation); unit: log ratio
Arm/Group | Pem + Carb or Cis (Non-Squamous) | Ram + Pem + Carb or Cis (Non-Squamous) | Gem + Carb or Cis (Squamous) | Ram + Gem + Carb or Cis (Squamous)
Number analyzed (Participants) | 53 | 58 | 50 | 53
log ratio | -0.2 (0.23) | -0.2 (0.22) | -0.3 (0.31) | -0.4 (0.39)
Statistical Analysis 1: Comparison: Pem + Carb or Cis (Non-Squamous) vs Ram + Pem + Carb or Cis (Non-Squamous); Test type: Superiority or Other; p = 0.1571, t-test, 2 sided
Statistical Analysis 2: Comparison: Gem + Carb or Cis (Squamous) vs Ram + Gem + Carb or Cis (Squamous); Test type: Superiority or Other; p = 0.1597, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Baseline through Study Completion (Up To 3 Years).
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Pem + Carb or Cis (Non-Squamous) | Ram + Pem + Carb or Cis (Non-Squamous) | Gem + Carb or Cis (Squamous) | Ram + Gem + Carb or Cis (Squamous)
All-Cause Mortality (participants affected / at risk) | 51/69 | 55/67 | 55/63 | 56/71
Serious Adverse Events (participants affected / at risk) | 38/69 | 44/67 | 29/63 | 39/71
Other Adverse Events (participants affected / at risk) | 67/69 | 66/67 | 62/63 | 71/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pem + Carb or Cis (Non-Squamous) (N=69) | Ram + Pem + Carb or Cis (Non-Squamous) (N=67) | Gem + Carb or Cis (Squamous) (N=63) | Ram + Gem + Carb or Cis (Squamous) (N=71)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 5 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 4 (5) | 2 (2) | 8 (10)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (5) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 5 (6) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (2) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 6 (8) | 1 (1) | 6 (7) | 7 (8)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Drug administration error (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 3 (4) | 2 (3) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Radiation mucositis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Underdose (Injury, poisoning and procedural complications) | 2 (2) | 4 (11) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 4 (5) | 1 (1) | 3 (3)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (3) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Air embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Embolism (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pem + Carb or Cis (Non-Squamous) (N=69) | Ram + Pem + Carb or Cis (Non-Squamous) (N=67) | Gem + Carb or Cis (Squamous) (N=63) | Ram + Gem + Carb or Cis (Squamous) (N=71)
Anaemia (Blood and lymphatic system disorders) | 37 (103) | 32 (95) | 40 (94) | 38 (111)
Leukopenia (Blood and lymphatic system disorders) | 4 (14) | 8 (20) | 10 (23) | 10 (36)
Neutropenia (Blood and lymphatic system disorders) | 17 (42) | 22 (70) | 35 (94) | 52 (152)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (48) | 22 (72) | 27 (73) | 36 (128)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Tachycardia (Cardiac disorders) | 4 (4) | 2 (2) | 4 (4) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 5 (7) | 3 (3) | 1 (1)
Lacrimation increased (Eye disorders) | 10 (10) | 8 (10) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 6 (8) | 4 (6) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (9) | 12 (17) | 3 (4) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (4) | 5 (6) | 4 (5)
Constipation (Gastrointestinal disorders) | 21 (29) | 19 (27) | 21 (28) | 18 (29)
Diarrhoea (Gastrointestinal disorders) | 19 (28) | 19 (23) | 12 (14) | 9 (12)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (6) | 6 (8) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 5 (7) | 4 (4) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1) | 4 (4)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 4 (6) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 39 (71) | 35 (65) | 36 (51) | 27 (44)
Stomatitis (Gastrointestinal disorders) | 6 (6) | 9 (13) | 6 (9) | 3 (3)
Vomiting (Gastrointestinal disorders) | 24 (34) | 22 (35) | 12 (15) | 18 (23)
Asthenia (General disorders) | 2 (2) | 8 (12) | 7 (10) | 5 (8)
Chills (General disorders) | 5 (5) | 1 (1) | 2 (2) | 5 (6)
Fatigue (General disorders) | 43 (85) | 44 (97) | 34 (62) | 39 (79)
Infusion site pain (General disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Mucosal inflammation (General disorders) | 6 (11) | 8 (14) | 5 (5) | 3 (3)
Non-cardiac chest pain (General disorders) | 3 (3) | 4 (11) | 4 (4) | 4 (4)
Oedema peripheral (General disorders) | 16 (19) | 17 (23) | 10 (12) | 14 (23)
Pyrexia (General disorders) | 12 (19) | 8 (9) | 6 (7) | 6 (8)
Nasopharyngitis (Infections and infestations) | 4 (8) | 2 (3) | 3 (4) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2) | 6 (6) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 8 (13) | 3 (3) | 4 (4)
Urinary tract infection (Infections and infestations) | 6 (15) | 7 (8) | 4 (6) | 3 (4)
Vulvovaginal mycotic infection (Infections and infestations) | 0/25 (0) | 1/33 (1) | 0/24 (0) | 1/16 (1)
Alanine aminotransferase increased (Investigations) | 7 (10) | 5 (10) | 6 (6) | 6 (17)
Aspartate aminotransferase increased (Investigations) | 4 (6) | 4 (8) | 6 (6) | 11 (24)
Blood alkaline phosphatase increased (Investigations) | 3 (6) | 1 (1) | 3 (5) | 7 (12)
Blood creatinine increased (Investigations) | 7 (8) | 6 (7) | 3 (3) | 4 (6)
Neutrophil count decreased (Investigations) | 7 (16) | 3 (3) | 3 (10) | 6 (9)
Platelet count decreased (Investigations) | 4 (7) | 3 (10) | 2 (3) | 7 (31)
Weight decreased (Investigations) | 11 (15) | 12 (17) | 4 (5) | 12 (16)
White blood cell count decreased (Investigations) | 5 (6) | 4 (8) | 5 (10) | 5 (15)
Decreased appetite (Metabolism and nutrition disorders) | 18 (27) | 20 (30) | 15 (17) | 24 (35)
Dehydration (Metabolism and nutrition disorders) | 12 (12) | 6 (6) | 5 (5) | 9 (9)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (12) | 3 (7) | 7 (9) | 6 (12)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 (12) | 1 (1) | 2 (3) | 10 (23)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 3 (3) | 6 (18)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (9) | 8 (9) | 8 (13) | 9 (14)
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 (15) | 10 (12) | 17 (23) | 14 (30)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (10) | 5 (11) | 5 (5) | 8 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (10) | 11 (16) | 5 (8) | 7 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (18) | 14 (21) | 9 (10) | 10 (14)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 3 (4) | 5 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 2 (2) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 8 (10) | 4 (5) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (11) | 3 (3) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (6) | 1 (1) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (9) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 13 (18) | 8 (8) | 6 (7) | 4 (4)
Dysgeusia (Nervous system disorders) | 6 (10) | 12 (16) | 8 (10) | 7 (7)
Headache (Nervous system disorders) | 8 (12) | 19 (33) | 5 (6) | 14 (20)
Hypoaesthesia (Nervous system disorders) | 4 (8) | 3 (6) | 1 (1) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 3 (4) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 4 (8) | 3 (5) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 4 (4) | 6 (6) | 4 (4) | 1 (1)
Depression (Psychiatric disorders) | 6 (7) | 5 (5) | 1 (1) | 5 (5)
Insomnia (Psychiatric disorders) | 10 (10) | 15 (15) | 7 (7) | 5 (5)
Proteinuria (Renal and urinary disorders) | 3 (3) | 3 (6) | 1 (1) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (18) | 13 (15) | 9 (9) | 14 (21)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (4) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (24) | 17 (29) | 11 (19) | 10 (19)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 4 (5) | 3 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 17 (36) | 6 (6) | 12 (17)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (3) | 4 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (10) | 3 (3) | 4 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 8 (9) | 6 (10)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7) | 1 (1) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 9 (9) | 8 (8) | 5 (5)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4) | 4 (4) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 4 (5) | 3 (4)
Hypertension (Vascular disorders) | 4 (5) | 12 (15) | 3 (4) | 8 (16)
Hypotension (Vascular disorders) | 3 (3) | 5 (7) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.